CLINICAL TRIAL: NCT02199444
Title: Effect of Sevelamer on P-cresol Levels in CKD
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Eleonora Riccio, MD, Federico II University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P-C Sev
Record Dates: First submitted 2014-07-22; First posted 2014-07-24 (Estimated); Last update posted 2015-02-18 (Estimated); Status verified 2014-09

CONDITIONS: Chronic Kidney Disease Stage 3-5
MeSH Terms: interventions — Sevelamer

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Sevelamer (Experimental): The dose of Sev was 2400 mg (800 mg three times a day) in all patients.
  Interventions: Drug: Sevelamer
- Placebo (Placebo Comparator): The patients received placebo three times a day
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sevelamer — The dose of Sev was 2400 mg (800 mg three times a day) in all patients.
  Arms: Sevelamer
Drug: Placebo
  Arms: Placebo

SUMMARY:
The accumulation of p-cresol, a product of the metabolism of aromatic aminoacid operated by resident intestinal bacteria increases the cardiovascular risk of chronic kidney disease (CKD) patients. Therefore, therapeutic strategies to reduce plasma p-cresol levels are highly demanded. It has been reported that the phosphate binder sevelamer sequesters p-cresol in vitro, while in vivo studies on dialysis patients showed controversial results. Aim of our study was to evaluate the effect of sevelamer on p-cresol levels in CKD patients.

ELIGIBILITY:
Inclusion Criteria:

* age >18 years,
* CKD stage 3-5

Exclusion Criteria:

* Existing or previous treatment within the last 1 year with a phosphate binder;
* hyperphosphatemia (>5.6 mg/dL);
* hypophosphatemia (<2.5 mg/dL);
* malnutrition,
* malignant neoplasms,
* current history of gastrointestinal and/or endocrine diseases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2014-06; Primary Completion 2015-05 (Estimated)

PRIMARY OUTCOMES:
Effect on p-creol levels | 3 months
  The p-cresol levels will be evaluated in plasma samples withdrawn after 1, 2 and 3 months of therapy.

CONTACTS AND LOCATIONS:
Locations (1):
- federico II university, department of nephrology, Naples, Italy, Italy

REFERENCES:
- [Derived] Natale P, Green SC, Ruospo M, Craig JC, Vecchio M, Elder GJ, Strippoli GF. Phosphate binders for preventing and treating chronic kidney disease-mineral and bone disorder (CKD-MBD). Cochrane Database Syst Rev. 2025 Jun 27;6(6):CD006023. doi: 10.1002/14651858.CD006023.pub4. PMID 40576086